CLINICAL TRIAL: NCT04648657
Title: Lung Ultrasound for Diagnosis of Lung Overdistension in Acute Hypoxaemic Respiratory Failure
Brief Title: Lung Ultrasound, PEEP and Overdistension (LUPO)
Acronym: LUPO
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Paolo Persona, principal investigator, University of Padova
Other Study IDs: 0021712
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Hypoxic Respiratory Failure
Keywords: lung ultrasound; lung overdistention; electric impedance tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- acute hypoxemic respiratory failure patients: Mechanically ventilated patients with acute hypoxemic respiratory failure (AHRF) with P/F ratio < 300 with at least PEEP 5 cmH2O)
  Interventions: Device: Lung Ultrasound; Device: Electric impedance tomography

INTERVENTIONS:
Device: Lung Ultrasound — Echography of Lungs based on artifacts study
  Other Names: LUS
Device: Electric impedance tomography — Low alternating electrical currents (usually <5 milliampere at 50-80 kHz) applied through different pair of electrodes on thorax
  Other Names: EIT

SUMMARY:
The investigators suppose that lung sliding could be reduced in the same lung region moving from less ventilated to overinflated condition. This is supported by theoretical arguments by some authors but so far it has not been demonstrated.

The investigators suppose that speckle tracking applied to LUS is able to demonstrate a reduction or abolition in pleural sliding when lung tissue is overinflated by higher PEEP after lung recruitment maneuver. The overinflation is diagnosed by Electric Impedance Tomography (EIT) and mechanical respiratory measurements (reduction in compliance as ratio between tidal volume over difference between plateau pressure and PEEP) and localized by EIT.

DETAILED DESCRIPTION:
Lung ultrasonography (LUS) is a rapid, easy and non-invasive bedside tool for the detection of specific ultrasound patterns, associated with several pulmonary and pleural disorders. The main limitation of studies assessing lung recruitability and lung monitoring during mechanical ventilation is the lack of detection of lung overinflation: the A pattern doesn't change if the lung tissue is completely re-aerated or is overinflated. Considering this, the investigators could not use LUS to guide lung recruitment due to the risk of lung damage. Speckle tracking echocardiography is a gray-scale based technique used for quantification of myocardial strain to provide a quantitative, objective measure of left ventricle (LV) systolic function.

The investigators suppose that lung sliding could be reduced in the same lung region moving from less ventilated to overinflated condition. This is supported by theoretical arguments by some authors but so far it has not been demonstrated.

The investigators suppose that speckle tracking is able to demonstrate a reduction or abolition in pleural sliding when lung tissue is overinflated by higher PEEP after lung recruitment maneuver. The overinflation is diagnosed by EIT and mechanical respiratory measurements (reduction in compliance as ratio between tidal volume over difference between plateau pressure and PEEP) and localized by EIT.

Primary endpoint: agreement between LUS and EIT to diagnose lung overdistension in Acute Hypoxaemic Respiratory failure patients during a PEEP trial.

Patients are ventilated in pressure controlled mode with a tidal volume of 6 mL/kg predicted body weight (PBW), respiratory rate (RR) is maintained as set per clinical management, I:E = 1:2, PEEP level is set at 5 cmH2O and inspiratory fraction of O2 (FiO2) at 100% before starting the protocol.

To check the presence of areas with reduced or absent pleural sliding not depending on overdistention, and to exclude absence of lung pulse due to pneumothorax, a basal LUS examination is performed before recruiting manoeuvre (RM): the ultrasound linear probe (12 megahertz, GE) is positioned parallel into the 4th-5th right intercostal space next to the sternal margin for the first acquisition; then other two acquisitions along the intercostal space from the medial part to the lateral side of the thorax are recorded; the procedure is repeated on the left side resulting in a final acquisition of 3 ultrasound clips of 10 seconds for each hemithorax. If the presence of pneumothorax is suspected or diagnosed (absence of lung pulse), the patient is excluded from the study according to exclusion criteria.

Then at the same level, marked with a dermographic pen, the EIT belt is positioned and a basal assessment of lung impedance is recorded.

After that a 40x40 RM is performed, setting a PEEP of 40 cmH2O for 40 seconds on continuous positive airway pressure mode mode. If hemodynamic instability or decrease in oxygen saturation occurs during the maneuver, RM is interrupted and previous ventilator settings restored until stability is obtained and the patient discharged from the protocol. If the presence of pneumothorax is suspected or diagnosed (absence of lung pulse), the patient is excluded from the study according to exclusion criteria and clinically managed.

Ventilation is then set again in volume controlled mode with a tidal volume of 6 ml/kg and a PEEP set to reach a maximum plateau pressure of 30 cmH20. I:E ratio and RR are left unchanged.

A decremental PEEP trial is performed reducing PEEP value of 2 cmH2O, static compliance is calculated with an inspiratory pause of 3 seconds just before PEEP modification, and a registration of EIT is acquired for each PEEP level. The PEEP trial starts with the maximum PEEP level (PEEPmax, which is 30 cmH2O minus the pressure generated by 6 ml/kg of tidal volume) and stops at 2 cmH2O less than the best PEEP (PEEPmin), identified according to the static compliance value.

At the same time ultrasound linear probe is transversely set 1 cm above or below the EIT belt and clips recorded at each PEEP level as described above (Fig.2). A total of 6 LUS clips for each level of PEEP is recorded.

Once best PEEP is identified, LUS clips are encoded stored on an external memory stick.

EIT images

Ultrasound setting pre-defined are fixed. Clips are analyzed using GE software and longitudinal speckle tracking applied for each pleural clip. A-lines are numbered per clip Measurements Maximal strain, strain rate and time to peak are calculated and stored by a second investigator blinded to respiratory maneuvers. Differences between parameters calculated on basal and on PEEP trial clips are analyzed.

EIT session is analyzed by dedicated software and lung impedance assessed; each LUS clip is matched with correspondent part of EIT image considered two Region of Interest on the upper part of each hemithorax.

Intra-observer variability on speckle-tracking is assessed by intra-class coefficient correlation; correlation between speckle tracking values and PEEP level is assessed by Spearman correlation test; receiving operating characteristic (ROC) curve (Youden's index) is calculated to predict the accuracy of speckle tracking for predicting hyperinflation. EIT and LUS clips are compared with Cohen's K.

A-lines are numbered at different level of PEEP to investigate if the number of A-lines could be related to lung overdistention

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* BMI < 35 kg/m2

Exclusion Criteria:

* Presence or history of pneumothorax, absence of lung pulse
* Pregnancy
* Patients with Pressure arterial O2/FiO2 (PaO2/FiO2) < 100 mmHg with at least 5 cmH2O of PEEP
* Pacemaker and/or internal cardiac defibrillator
* Hemodynamic parameters: systolic blood pressure <100 mmHg and >180 mmHg, or if systolic blood pressure is between 100-180 mmHg on high dose of IV continuous infusion of norepinephrine (>0,2 μg/kg/min), or dobutamine (>5 μg/kg/min ), or dopamine (>5 μg/kg/min), or epinephrine (>0,1 μg/kg/min)
* Hemodynamic instability (systolic blood pressure < 70 mmHg, heart rate increase to >140 bpm or decrease to <60 bpm, appearance of cardiac arrhythmias, (peripheral saturation O2 (SpO2) decrease to < 88%) during RM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated patients with acute hypoxemic respiratory failure (AHRF) or acute respiratory distress syndrome (ARDS) according to the Berlin definition (P/F ratio 100-300 with at least PEEP 5 cmH2O)
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
agreement between LUS+Speckle tracking and EIT in diagnosis of lung overdistension | 5 months
  LUS with speckle tracking applied and EIT are able to diagnose lung overdistension in the same lung zone

SECONDARY OUTCOMES:
quantification of lung sliding by speckle tracking at different levels of PEEP | 5 months
  Speckle tracking applied to LUS is able to quantify lung sliding at different PEEP levels
correlation between number of A-lines and lung overdistention | 5 months
  the number of A-lines per clip at different level of PEEP is related to the lung overdistention diagnosed by EIT

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Navalesi, MD, Study Chair — University of Padova
Locations (1):
- Azienda Ospedaliera Università di Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bikker IG, Leonhardt S, Reis Miranda D, Bakker J, Gommers D. Bedside measurement of changes in lung impedance to monitor alveolar ventilation in dependent and non-dependent parts by electrical impedance tomography during a positive end-expiratory pressure trial in mechanically ventilated intensive care unit patients. Crit Care. 2010;14(3):R100. doi: 10.1186/cc9036. Epub 2010 May 30. PMID 20509966
- [Background] Duclos G, Bobbia X, Markarian T, Muller L, Cheyssac C, Castillon S, Resseguier N, Boussuges A, Volpicelli G, Leone M, Zieleskiewicz L. Speckle tracking quantification of lung sliding for the diagnosis of pneumothorax: a multicentric observational study. Intensive Care Med. 2019 Sep;45(9):1212-1218. doi: 10.1007/s00134-019-05710-1. Epub 2019 Jul 29. PMID 31359081
- [Background] Uematsu M. Speckle tracking echocardiography - Quo Vadis? Circ J. 2015;79(4):735-41. doi: 10.1253/circj.CJ-15-0049. Epub 2015 Mar 13. PMID 25766514
- [Background] Hickling KG. Best compliance during a decremental, but not incremental, positive end-expiratory pressure trial is related to open-lung positive end-expiratory pressure: a mathematical model of acute respiratory distress syndrome lungs. Am J Respir Crit Care Med. 2001 Jan;163(1):69-78. doi: 10.1164/ajrccm.163.1.9905084. PMID 11208628
- [Background] Adler A, Amyot R, Guardo R, Bates JH, Berthiaume Y. Monitoring changes in lung air and liquid volumes with electrical impedance tomography. J Appl Physiol (1985). 1997 Nov;83(5):1762-7. doi: 10.1152/jappl.1997.83.5.1762. PMID 9375349